CLINICAL TRIAL: NCT02341794
Title: Rosuvastatin Treatment for Intracranial Arterial Stenosis Based on Magnetic Resonance Angiography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tokyo Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2900
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Intracranial Arterial Diseases
Keywords: intracranial arterial disease; dyslipidemia; rosuvastatin
MeSH Terms: conditions — Intracranial Arterial Diseases; Dyslipidemias | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rosuvastatin (Experimental)
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin (5mg) will be orally administrated once daily. Dose of rosuvastatin will be adjusted to control serum LDL-c level under 1.8 mmol/L.

SUMMARY:
The purpose of this study is to investigate the effects of rosuvastatin treatment on degree of intracranial arterial stenosis.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects of rosuvastatin treatment on degree of intracranial arterial stenosis in two years. Dyslipidemia patients with intracranial arterial stenosis will be enrolled under informed consent in this study. Rosuvastatin (5mg) will be orally administered once daily. Dose of rosuvastatin will be adjusted to control serum LDL-c level under 1.8mmol/L. Primary outcome is the progression of intracranial stenosis on magnetic resonance angiography (MRA) after two years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between 30 and 80 years of age.
2. Patients with noncardioembolic ischemic stroke
3. Patients with intracranial arterial stenosis ≥50% in supraclinoid internal carotid artery, M1 portion of middle cerebral artery, A1 portion of anterior cerebral artery, P1 portion of posterior cerebral artery, or basilar artery.
4. LDL-C level is more than 100 mg/dl (2.6 mmol/L) or under treatment of dyslipidemia
5. Patients taking clopidogrel as antiplatelet therapy when providing informed consent
6. Patients considered to be able to visit the study site
7. Patients who provided written informed consent

Exclusion Criteria:

1. Any haemorrhagic stroke or haemorrhagic infarction
2. Familial hypercholesterolemia
3. Patients with uncontrolled angina pectoris or congestive heart failure
4. Patients with severe liver or renal dysfunction
5. Patients with a malignant tumor requiring treatment
6. Patients with uncontrolled diabetes mellitus
7. Patients with secondary dyslipidemia (due to corticosteroid etc)
8. Patients with a history of myopathy
9. Patients considered by the investigator to be unsuitable for participating in this study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Progression of intracranial arterial stenosis after two years | 6 months, 1 year and 2 years

SECONDARY OUTCOMES:
Any stroke (ischemic stroke, intracerebral haemorrhage, subarachnoid haemorrhage) | 6 months, 1 year and 2 years
Ischemic stroke or transient ischemic attack | 6 months, 1 year and 2 years
Intracerebral haemorrhage or subarachnoid haemorrhage | 6 months, 1 year and 2 years
Death from any cause | 6 months, 1 year and 2 years
Cardiovascular events (ischemic stork, cardiac infarction, and other vascular events | 6 months, 1 year and 2 years
The change of percentage in LDL-C from baseline | 6 months, 1 year and 2 years
The change in HDL-C level from baseline | 6 months, 1 year and 2 years
Intracranial haemorrhage | 6 months, 1 year and 2 years
Number of cerebral microbleeds on MRI | 6 months, 1 year and 2 years
Carotid intima-media thickness | 6 months, 1 year and 2 years
Ankle brachial index | 6 months, 1 year and 2 years
Brachial-ankle pulse wave velocity | 6 months, 1 year and 2 years
Adverse events and adverse drug reactions | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hitoshi Aizawa, MD, PhD, Principal Investigator — Tokyo Medical University
Locations (1):
- Tokyo Medical University, Shinjuku-ku, Tokyo, Japan